CLINICAL TRIAL: NCT03637543
Title: A Phase 2 Study of Nivolumab in Patients With High-Risk Biochemically Recurrent Prostate Cancer
Brief Title: Nivolumab in Patients With High-Risk Biochemically Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David J. Einstein, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-249
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PD-L1 Positive (Experimental): -Nivolumab will be given on day 1 of a 28-day cycle intravenously
  Interventions: Drug: Nivolumab
- PD-L1 Negative (Experimental): -Nivolumab will be given on day 1 of a 28-day cycle intravenously
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is an antibody inhibitor of the programmed death-1 (PD-1) pathway. By blocking PD-1, this medication may allow the immune system to recognize and fight cancer
  Other Names: Opdivo

SUMMARY:
This research study is studying an immune-based cancer drug as a possible treatment for prostate cancer.

The drug involved in this study is:

-Nivolumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved nivolumab for this specific disease but it has been approved for other uses. Nivolumab is an antibody inhibitor of the programmed death-1 (PD-1) pathway. By blocking PD-1, this medication may allow the immune system to recognize and fight cancer.

In this research study, the investigators are investigating whether nivolumab has any activity in patients who have a rising PSA (prostate specific antigen) after previously undergoing surgery or radiation for prostate cancer. Although nivolumab was previously not found to have significant effect in advanced prostate cancer after all other therapies had failed, based on new research, the investigators are testing whether nivolumab could have a greater effect earlier in the disease course and before patients receive hormone therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed an informed-consent form indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.
* Patients must have a history of prostate adenocarcinoma (adenocarcinoma must be the primary histology; secondary components of variant histologies are acceptable) confirmed on biopsy and treated with primary radical prostatectomy (RP) or definitive radiation (RT). Prior salvage RT is acceptable.
* Patients must have experienced biochemical recurrence (BCR) plus have minimum PSA values noted below:

  * Following primary RP: Any detectable rising PSA after RP (or after salvage RT if performed), minimum PSA 1.0 at time of screening
  * Following primary RT: PSA rise to ≥2 ng/mL above the nadir
  * No evidence of metastases on conventional imaging (CT or MRI plus bone scan)
* PSA doubling time (PSADT) <10 months --PSADT: calculated as per Prostate Cancer Working Group 3 (PCWG3) and the Memorial Sloan Kettering Cancer Center calculator: (https://www.mskcc.org/nomograms/prostate/psa_doubling_time)

With linear regression model of normal logarithm of PSA and time, based on:

* At least 3 consecutive PSA values with each value ≥0.2 ng/mL
* Interval between first and last PSA values is ≥8 weeks but ≤12 months.

  -Archival tissue is mandatory, either prostatectomy specimen or (in patients who received primary RT) diagnostic core biopsies. Patients must consent to next-generation sequencing performed on this tissue.
* If diagnostic core biopsies are only available tissue, at least 3 cores must be involved by tumor

  * Easteron Cooperative Oncology Group (ECOG) performance status 0-1
  * Age ≥18 years
  * Adequate organ and marrow function:
  * System Laboratory Value
* Hematological
* White blood cell (WBC) ≥ 2000/µL
* Absolute Neutrophil Count (ANC) ≥ 1500/μL
* Platelets (Plt) ≥ 100 x103/μL
* Hemoglobin (Hgb) > 9.0 g/dL (with or without transfusion)

  -Renal
* Serum Creatinine ≤ 2 x ULN
* Hepatic
* Bilirubin1 ≤ 1.5× upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 3 × ULN
* Alanine aminotransferase (ALT) ≤ 3 × ULN

  * Except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL
  * Baseline testosterone ≥100 ng/dL
  * Recovery from acute toxicity related to prior therapy, including surgery and radiation, or no treatment-related toxicity ≥ grade 2.
  * History of prior malignancy or concurrent separate malignancy is not an exclusion criterion so long as the non-prostate malignancy is stable and does not require any treatment.
  * Able to understand and sign informed consent and adhere to study procedures.
  * Male patients whose female partners are of reproductive potential must agree to use a contraception during the trial period

Exclusion Criteria:

* Current use of ADT or plan to initiate ADT during trial period
* Major surgery or radiation therapy within 14 days of starting study treatment
* Subjects with active autoimmune disease. Patients with a history of autoimmune disease that has not required systemic immunosuppressive therapy or does not threaten vital organ function including central nervous system, heart, lungs, kidneys, skin, and gastrointestinal tract will be allowed.
* Known history of immune deficiencies or chronic viral infections including HIV, hepatitis B (HBV), and hepatitis C (HCV) (patients with prior therapy for HBV or HCV is permitted if viral clearance was documented).
* Concurrent medical condition requiring use of systemic corticosteroids with prednisone >10 mg per day or equivalent. Use of inhaled, nasal, and topical steroids (applied to small body areas) is allowed.
* Current use (within past 4 weeks) of other prohibited medications including anti-cancer therapies, hormonal therapies, 5-alpha reductase inhibitors, and alternative medications known to alter PSA (e.g. phytoestrogens and saw palmetto).
* Prior treatment with immune checkpoint inhibitors. (Prior cancer vaccines are allowed.)
* Serious intercurrent medical or psychiatric illness that, in the judgment of the investigator, would interfere with patient's ability to carry out the treatment program

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Control | 12 weeks
  Proportion of patients with high-risk biochemically-recurrent (BCR) prostate cancer (PCa) that experiences decline or stabilization in PSA (without symptomatic/radiographic progression) after 12 weeks of nivolumab treatment

SECONDARY OUTCOMES:
Maximal change in prostate specific antigen (PSA) during nivolumab treatment | 2 years
Best PSA response during nivolumab treatment as an absolute change relative to baseline | 2 years
Change in PSA doubling time (PSADT) at end-of-study relative to baseline | 2 years
Time from enrollment to development of radiographic metastatic disease | 2 years
Time from enrollment to initiation of androgen deprivation therapy (ADT) | 2 years
Treatment-related adverse events as assessed by CTCAE v5.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Einstein, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - DFCI South Shore, South Weymouth, Massachusetts
  - DFCI Londonderry, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: No